CLINICAL TRIAL: NCT05043376
Title: Study to Investigate the Treatment Effect of Probiotic Streptococcus Salivarius K12 in Hospitalised Patients (Non-ICU) With COVID-19
Brief Title: Study to Investigate the Treatment Benefits of Probiotic Streptococcus Salivarius K12 for Hospitalised Patients (Non-ICU) With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, somia iqtadar, Associate Professor of Medicine, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 625/RC/KEMU/07.09.2021
Record Dates: First submitted 2021-09-11; First posted 2021-09-14 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): In this arm patients will receive the standard COVID-19 care as per the hospital guidelines.
  Interventions: Drug: Standard of care
- BLIS K12 (Experimental): In this arm patients will receive the BLIS K12 as add-on to the standard COVID-19 care
  Interventions: Drug: Standard of care; Dietary Supplement: BLIS K12

INTERVENTIONS:
Drug: Standard of care — Standard COVID-19 care as per the hospital guidelines
Dietary Supplement: BLIS K12 — Daily 2 oral BLIS K12 tablets for up to 14 days.
  Arms: BLIS K12

SUMMARY:
This is a randomised, open-label and controlled clinical trial aimed to investigate the adjuvant treatment benefits of probiotic Streptococcus salivarius K12 in hospitalised mild-to-moderate patients with COVID-19 disease.

DETAILED DESCRIPTION:
Boosting the immunity and maintaining a healthy and balanced microflora at oropharyngeal environment of people through probiotics supplementation has been proposed as a possible strategy to protect human host from respiratory tract infections. A slow-dissolved oropharyngeal probiotic formula containing S. salivarius K12 has been clinically demonstrated to improve the upper respiratory tract microbiota protecting the host from pathogenic bacteria, fungi, and viruses, thereby reducing the incidence of viral respiratory tract infections and bacterial co-infections. S. salivarius K12 has been proposed as a promising agent for prophylactic or probiotic treatments to protect individuals during the outbreak of seasonal or emerging respiratory infection diseases.

S. salivarius K12 strain, commonly known as BLIS K12, is a highly safe, and extensively-studied probiotic that resides in the oral cavity. BLIS K12 has a solid scienctific rationale for helping to prevent streptococcal pharyngitis and/or tonsillitis, ear infections (otitis media) and to help treat halitosis. It is a specific strain of Streptococcus Salivarius, which secretes powerful anti-microbial molecule called Bacteriocin-Like-Inhibitory Substances (BLIS). The ingredient is believed to support healthy bacteria in the mouth for long-term fresh breath and immune support.

It is proposed that the oral administration of the strain K12 to hospitalized COVID-19 patients (not already in ICU) receiving supplementary oxygen (not invasive oxygen theraphy) to exploit the "ventilation" and helping S. salivarius (K12) to move from the mouth (it is an oral colonizer) to the lungs, colonizing them. The idea is that the lung presence of K12 could strategically reduce the lung and immune capability to release pro-inflammatory cytokines, thus preventing excessive lung inflammation, and the need to proceed to ICU and death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (both sexes)
* Hospitalized confirmed (RT-PCR) COVID-19 patients (not already in ICU) admitted for treatment of COVID-19 and not receiving mechanical ventilatory support
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with proven hypersensitivity or allergic reaction to the tested formula
* Patients who decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Recovery and live discharge | From day 1 to day 14
  Number of patients with clinical improvement

SECONDARY OUTCOMES:
Hospitalisation days | From day 1 to day 14
  The effect of K12 treatment in reducing the hospitalisation days
Effect on inflammatory markers | From day 1 to day 14
  Numbers of patients with improvement in the inflammatory markers
ICU transfer | From day 1 to day 14
  Reduction in the rate of ICU transfer

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No